CLINICAL TRIAL: NCT03414905
Title: Management of Malignant Pleural Effusions Using an Indwelling Tunneled Pleural Catheter and Non-Vacuum Collection System
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 201708040
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Aspira Catheter & Drainage System: * Participants will have standard of care ultrasound and placement of the Aspira Catheter and Drainage System on Day 1
  * The removal of the Aspira Catheter and Drainage System will be dependent upon future ultrasound assessment and fluid output
  Interventions: Device: Aspira Catheter; Procedure: Ultrasound

INTERVENTIONS:
Device: Aspira Catheter — * 15.5Fr catheter
  * Standard of care
  Other Names: Aspira Catheter and Drainage System
Procedure: Ultrasound — Standard of care

SUMMARY:
In this study, the investigators will collect data on patients who are using the Aspira system as part of their clinical care for the management of recurrent pleural effusion. Data will be collected on patient demographics, placement of the pleural catheter, palliation of dyspnea, complication rates, and rates of spontaneous pleurodesis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years of age, inclusive
* Subject has a symptomatic malignant pleural effusion requiring intervention. For an effusion to be defined as malignant, at least one of the following must be true

  * There is cytological confirmation of pleural malignancy
  * The effusion is an exudate (per Light's criteria Pleural fluid protein/Serum protein >0.5, Pleural fluid LDH/Serum LDH >0.6, or Pleural fluid LDH >2/3 the upper limit of normal) in the context of histocytologically proven malignancy elsewhere, with no other clear cause for fluid identified
* Subject is able to provide informed consent
* Subject has sufficient pleural fluid to allow safe insertion of an indwelling tunneled pleural catheter as determined by the PI
* Subject is able to perform home drainage of the pleural effusion or has sufficient resources (family member, caregiver, home health).

Exclusion Criteria:

* Subject is pregnant
* Subject has evidence, in the opinion of the PI, of either ongoing systemic or pleural infection
* Subjects with uncorrected coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants will be seen at Washington University School of Medicine.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Relief of dyspnea as measured using the Visual Analog Scale for Dyspnea (VAS-Dyspnea) | Through 2 weeks following catheter insertion
  * This will be determined based on the difference between the VAS-Dyspnea score on the day of catheter insertion prior to catheter insertion compared with the VAS-Dyspnea score on the 2 week follow up visit
  * The scale presents the question "how much shortness of breath are you having right now?" with a straight line. At one end it states "no shortness of breath" and the other end is "shortness of breath as bad as can be". The participant will mark the line on how they feel
  * No shortness is breath is 0% score and shortness of breath as bad as can be is 100% score

SECONDARY OUTCOMES:
Rate of infection | 1 year
  -Defined as the isolation of any bacteria within a pleural fluid specimen drawn for clinical purposes
Rate of spontaneous pleurodesis | 1 year
  -Defined as pleural fluid drainage less than 75ml every other day for three consecutive drainage sessions

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Chen, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu